CLINICAL TRIAL: NCT02084264
Title: Multicenter, Prospective, Partially Randomized, Controlled Trial of Robotic-guided vs. Freehand Corrective Surgery for Pediatric Scoliosis
Brief Title: Robotic vs. Freehand Corrective Surgery for Pediatric Scoliosis
Acronym: PEDSCOLI
Status: Terminated | Type: Observational
Why Stopped: Administrative
Sponsor: Mazor Robotics (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN108
Record Dates: First submitted 2014-03-09; First posted 2014-03-11 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Scoliosis
Keywords: Adolescent Idiopathic Scoliosis; Pediatric Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arm 1: Robotic-guided, open approach: Robotic-guided, open approach
- Arm 2: control arm- non-robotic, open approach: control arm- non-robotic, open approach°

SUMMARY:
To compare the accuracy and feasibility, curvature correction and clinical outcomes of pedicle screw instrumentation with versus without robotic guidance, in pediatric and adolescent scoliosis patients

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric/adolescent patients (age 10 to 21 years), undergoing a primary surgery for the correction of a scoliotic curve of 40 degrees or greater
2. Patient capable of complying with study requirements
3. Signed informed consent by patient

Exclusion Criteria:

1. Scheuermann's disease
2. Infection or malignancy
3. Primary abnormalities of bones (e.g. osteogenesis imperfecta)
4. Primary muscle diseases, such as muscular dystrophy
5. Neurologic diseases (e.g. Charcot-Marie Tooth, Guillain-Barre syndrome, cerebral palsy, spina bifida, or neurofibroma)
6. Spinal cord abnormalities with any neurologic symptoms or signs
7. Spinal cord lesions requiring neurosurgical interventions, such as hydromyelia
8. Patients who have participated in a research study involving an investigational product in the 12 weeks prior to surgery
9. Patients requiring anterior release or instrumentation
10. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study.
11. Pregnancy
12. Patient cannot follow study protocol, for any reason
13. Patient cannot or will not sign informed consent

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric/adolescent patients (age 21 years and younger) undergoing a primary surgery for the correction of a scoliotic curve of 40 degrees or greater
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2014-10; Primary Completion 2019-07-08 (Actual); Study Completion 2019-07-08 (Actual)

PRIMARY OUTCOMES:
Revision surgeries | 1 year post-surgery
  All cause revisions, including medical and surgical complications.

SECONDARY OUTCOMES:
Clinical performance of instrumentation technique | Day of surgery
  instrumentation time per screw, total surgery time, excluding: exposure and closure time, Surgeon-specific surgical techniques that impact surgery time
Neuromonitoring events | Day of surgery
Hypoplastic pedicles | Day of surgery
  <4 mm in diameter
Improvement of radiographic and health-related quality of life metrics | up to 10 years post-operative
  post-operative radiographs and SRS22 questionnaire
Length of convalescence | within 2 years of surgery
  Length of hospital stay, destination at discharge, time to return to normal activities
Clinical Outcomes as measured on plain radiographs | 2 years
  Curvature correction and shoulder balance
Radiation Exposure | Day of surgery
  Reading of exposure in seconds (and KvP, if available) from C-arm or other imaging system used in the operating room.
Ratio of executed vs. planned screws | Day of surgery
  Number of screws planned to be robotically inserted and manually inserted instead, and cause.
Pedicle screw instrumentation accuracy | Within 1 year of surgery, if indicated by surgeon and clinically necessary
  Accuracy will be quantified in millimeters and scored using the Gertzbein-Robbins classification, based on post-operative CTs that are clinically necessary for the management of the patient.
Surgical complications | Within first year from day of surgery
  Implant-related durotomy, infection requiring surgery, excessive blood loss, air emboli, new neural deficits, implant failure

CONTACTS AND LOCATIONS:
Overall Officials: Doron Dinstein, MD, Study Director — Mazor Robotics
Locations (4):
- United States (4):
  - Rady Children's Hospital- San Diego, San Diego, California
  - Florida Hospital for Children, Orlando, Florida
  - Children's Healtchare of Atlanta at Scottish Rite, Atlanta, Georgia
  - Geisinger Orthopaedic Institute, Danville, Pennsylvania

REFERENCES:
- [Background] Devito DP, Kaplan L, Dietl R, Pfeiffer M, Horne D, Silberstein B, Hardenbrook M, Kiriyanthan G, Barzilay Y, Bruskin A, Sackerer D, Alexandrovsky V, Stuer C, Burger R, Maeurer J, Donald GD, Schoenmayr R, Friedlander A, Knoller N, Schmieder K, Pechlivanis I, Kim IS, Meyer B, Shoham M. Clinical acceptance and accuracy assessment of spinal implants guided with SpineAssist surgical robot: retrospective study. Spine (Phila Pa 1976). 2010 Nov 15;35(24):2109-15. doi: 10.1097/BRS.0b013e3181d323ab. PMID 21079498